CLINICAL TRIAL: NCT04990154
Title: Effects of Intradialytic Exercise on Dialytic Parameters, Health-related Quality of Life, and Depression Status in Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Effects of Intradialytic Exercise on Health-related Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, CHIA-HUEI LIN, PhD, Associate professor, Tri-Service General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSGHIRB: 1-108-05-070
Record Dates: First submitted 2021-07-23; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Exercise
Keywords: intradialytic exercise; hemodialysis; health-related quality of life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A randomized, controlled trial with a two parallel-group design
Who Masked: Outcomes Assessor
Masking Description: outcome assessor was blinded to the group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group received a 12-week intradialytic exercise (supine lower-limb ergometer, 30 minutes/session, 3 sessions/week)
  Interventions: Behavioral: a 12-week intradialytic exercise
- control group (No Intervention): the control group maintained their usual lifestyles

INTERVENTIONS:
Behavioral: a 12-week intradialytic exercise — a 12-week intradialytic exercise (supine lower-limb ergometer, 30 minutes/session, 3 sessions/week)
  Arms: experimental group

SUMMARY:
This study aimed to evaluate the effects of intradialyic exercise on dialytic parameters, HRQL, and depression status in hemodialysis patients. A randomized controlled trial was conducted. Sixty-four participants were recruited using stratified random sampling and allocated with a 1:1 randomization ratio to either experimental group (EG, treated in odd weekdays, n = 32) or comparison group (CG, treated in even weekdays, n = 32). The EG received a 12-week intradialytic exercise, while the CG maintained usual lifestyles. Dialytic parameters, HRQL, and depression status were collected at baseline and at 12 weeks. The results indicated that there were no differences in changes of dialytic parameters from baseline between EG and CG. However, the EG had increased HRQL and reduced depression status at 12 weeks compared with the CG. A 12-week intradialytic exercise is safe, feasible and effective in improved HRQL and reduced depression status for hemodialysis patients.

DETAILED DESCRIPTION:
Exercise has been shown to be of fundamental importance in managing chronic diseases and improving health-related quality of life (HRQL) as well as psychological health. However, whether intradialyic exercise is safe and has positive impact on HRQL and depression status in hemodialysis patients requires further researches with diverse racial and cultural groups to clarify. This study aimed to evaluate the effects of intradialyic exercise on dialytic parameters, HRQL, and depression status in hemodialysis patients. A randomized controlled trial was conducted at a medical center in Northern Taiwan. Sixty-four participants from 112 eligible hemodialysis patients were recruited using stratified random sampling and allocated with a 1:1 randomization ratio to either experimental group (EG, treated in odd weekdays, n = 32) or comparison group (CG, treated in even weekdays, n = 32). The EG received a 12-week intradialytic exercise (supine lower-limb ergometer, 30 minutes/session, 3 sessions/week), while the CG maintained usual lifestyles. Dialytic parameters (serum chemistries, serum electrolytes, and estimated glomerular filtration rate), HRQL, and depression status were collected at baseline and at 12 weeks. The results indicated that there were no differences in changes of dialytic parameters from baseline between EG and CG. However, the EG had increased HRQL (ß = 22.6, p<.001) and reduced depression status (ß = -7.5, p = .02) at 12 weeks compared with the CG. A 12-week intradialytic exercise is safe, feasible and effective in improved HRQL and reduced depression status for hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* (1) ESRD patients on maintenance of hemodialysis; (2) aged 20 to 80 years; (3) able to speak and understand Mandarin; (4) had received regular treatment with hemodialysis (3 times/ week) for at least 6 months; (5) agreed to be randomized to one of the two groups.

Exclusion Criteria:

* lower limb disabilities, hospitalized patients, treatment with peritoneal dialysis, received hemodialysis less than 3 times/ week, a history of recent acute myocardial infarction, unstable angina, uncontrolled arrhythmia, acute stroke, hospitalization experience within 6 months, cancer, and diagnosed with mental illness, especially depression.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-05-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Dialytic parameters: red blood cell [count/ul] | Change from baseline red blood cell [count/ul] assessed by blood analysis at 12 weeks
  red blood cell [count/ul]
Dialytic parameters: hemoglobin [g/dl] | Change from baseline hemoglobin [g/dl] assessed by blood analysis at 12 weeks
  hemoglobin [g/dl]
Dialytic parameters: hematocrit [%] | Change from baseline hematocrit [%] assessed by blood analysis at 12 weeks
  hematocrit [%]
Dialytic parameters: mean corpuscular volume [fl] | Change from baseline mean corpuscular volume [fl] assessed by blood analysis at 12 weeks
  mean corpuscular volume [fl]
Dialytic parameters: albumin [g/dl] | Change from baseline albumin [g/dl] assessed by blood analysis at 12 weeks
  albumin [g/dl]
Dialytic parameters: GPT [IU/l] | Change from baseline [IU/l] assessed by blood analysis at 12 weeks
  GPT [IU/l]
Dialytic parameters: GOT [IU/l] | Change from baseline GOT [IU/l] assessed by blood analysis at 12 weeks
  GOT [IU/l]
Dialytic parameters: blood urea nitrogen [BUN, mg/dl] | Change from baseline blood urea nitrogen [BUN, mg/dl] assessed by blood analysis at 12 weeks
  blood urea nitrogen [BUN, mg/dl]
Dialytic parameters: creatinine [Cr, mg/dl]) | Change from baseline creatinine [Cr, mg/dl]) assessed by blood analysis at 12 weeks
  creatinine [Cr, mg/dl])
Dialytic parameters: sodium [Na, mEq/l] | Change from baseline sodium [Na, mEq/l] assessed by blood analysis at 12 weeks
  sodium [Na, mEq/l]
Dialytic parameters: potassium [K, mEq/l] | Change from baseline potassium [K, mEq/l] assessed by blood analysis at 12 weeks
  potassium [K, mEq/l]
Dialytic parameters: calcium [Ca, mg/dl] | Change from baseline calcium [Ca, mg/dl] assessed by blood analysis at 12 weeks
  calcium [Ca, mg/dl]
Dialytic parameters: phosphate [P, mg/dl] | Change from baseline phosphate [P, mg/dl] assessed by blood analysis at 12 weeks
  phosphate [P, mg/dl]
Dialytic parameters: IPTH [pg/ml] | Change from baseline IPTH [pg/ml] assessed by blood analysis at 12 weeks
  IPTH [pg/ml]
Dialytic parameters: estimated GFR [ml/min1.73m2]) | Change from baseline estimated GFR [ml/min1.73m2]) assessed by estimation based on serum creatinine at 12 weeks
  estimated GFR [ml/min1.73m2])
health-related quality of life assessed by the scale of SF-36 | Change from baseline health-related quality of life at 12 weeks
  self-reported health-related quality of life
depression status assessed by the scale of Beck Depression inventory | Change from baseline depression status at 12 weeks
  self-reported depression status

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Huei Lin, PhD, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Chia-Huei Lin, Taipei, Hawaii, Taiwan